CLINICAL TRIAL: NCT04516304
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Assess a Nutritional Supplement on Vasomotor Symptoms In Perimenopausal and Menopausal Women
Brief Title: A Nutritional Supplement on Vasomotor Symptoms in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmavite LLC (Industry)
Collaborators: Biofortis, Merieux NutriSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIO-1811
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Menopause
Keywords: menopause
MeSH Terms: interventions — Equol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: S-equol
- Experimental (Experimental): S-equol
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: S-equol

INTERVENTIONS:
Dietary Supplement: Placebo — 4 tablets/d (2 in the morning and 2 in the evening)
Dietary Supplement: S-equol — 4 tablets/d (2 in the morning and 2 in the evening), providing 10 mg S-equol total a day Other Names: •Equelle®

SUMMARY:
Vasomotor symptoms (VMS), such as flushes, sweating, and sleep disturbances, are experienced by up to 80% of women during the menopausal transition. Night sweats, which are hot flushes that occur at night, can be particularly bothersome in women and contribute to disturbed sleep. These symptoms occur mainly during the 1-3 years prior to menopause (late perimenopause) and early menopause (~4 years after menstruation ceases). Many women look to supplements for the management of menopausal symptoms. Soy isoflavones and their metabolites are one category of dietary supplements that have been extensively studied for the management of VMS. The most active soy isoflavone is S-equol, which is not found directly in soy, but rather is the metabolite that is produced by gut microflora from consumption of the soy isoflavone daidzein. However, only 20-30% of US women are actually able to produce S-equol from the consumption of daidzein. Equelle® is a currently available dietary supplement that has S-equol as its active component, which allows the delivery of the active soy isoflavone metabolite directly without dependence on the gut microflora metabolism. The intention of this study is to assess the effect of a product containing S-equol on the management of VMS in normally healthy women.

Condition or disease: Vasomotor Symptoms

Intervention/treatment:

Dietary Supplement: S-equol Dietary Supplement: Placebo

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, parallel study, which will include a screening visit (Visit 1; week -3), a 2-week run-in period for baseline determination and assessment of placebo response (Visit 2; week -2; and Visit 3; week -1), one baseline visit (Visit 4; week 0), and three test visits (Visits 5, 6, and 7; weeks 4, 8, and 12).

At Visit 1 (week -3), after subjects have provided informed consent, medical history will be reviewed, and clinic visit procedures will be performed, including assessments of prior/current medication/supplement use, evaluations of inclusion/exclusion criteria, and a last menses query. Fasting (10-14 h) blood samples will be collected for assessment of FSH and estradiol levels. The Soy Food Frequency Questionnaire will be administered and subjects will be instructed to maintain their habitual diets (with the exception of avoiding soy foods) and physical activity patterns throughout the study period. Additionally, subjects will be dispensed the Insomnia Severity Index Questionnaire (ISIQ) and the VMS Diary to assess insomnia and VMS, respectively.

At Visit 2 (week -2), eligible subjects will be instructed to start the run-in placebo product for two weeks. Subjects will be also instructed to continue daily recording in the VMS Diary. At Visit 3 (week -1), the VMS Diary will be collected/reviewed to assess response to the run-in placebo product. Subjects who continue to meet the inclusion/exclusion criteria will be allowed to continue with the study and will be dispensed a sleep tracking device to wear for sleep/wake pattern evaluation.

At Visit 4 (week 0), eligible subjects will be randomized to one of the study products (Active or Placebo) and instructed to consume with water for 12 weeks. Additionally, the Pittsburg Sleep Quality Index (PSQI), RAND-36 Questionnaire, Profile of Mood States (POMS), Day-to-Day Impact of Vaginal Aging Questionnaire (DIVQ), Chalder Fatigue Scale, and Menopause-Specific Quality of Life (MENQOL) Questionnaire will be administered. The VMS Diary and ISIQ will be collected and reviewed.

At Visits 5 and 6 (weeks 4 and 8), the VMS Diary and ISIQ will be collected/reviewed, and the PSQI and MENQOL will be administered. Subjects will return to the clinic prior to Visit 7 (week 12) to receive the sleep tracking device to wear for sleep/wake pattern evaluation one week (7 d) prior to Visit 7 (week 12).

At Visit 7 (week 12), the VMS Diary and ISIQ will be collected and reviewed. The PSQI, RAND-36, POMS, DIVQ, Chalder Fatigue Scale, and MENQOL will be administered and study product will be collected/reviewed, and compliance will be determined. Additionally, the sleep tracker will be collected, and data will be downloaded for evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a perimenopausal or menopausal female experiencing specific menopausal-related VMS.
2. Subject has a BMI of ≥18.5 to ≤38.0 kg/m2 at Visit 1 (week -3).
3. At screening visit (Visit 1; week -3), subject reports to have 4 or more moderate to severe hot flushes/night sweats during 24 h prior to the visit. At Visit 3 (week -1), subject has ≥25 moderate to severe hot flushes/night sweats per week for one week between Visit 2 and 3 (weeks -2 and -1). At Visit 4 (week 0), subject has an average ≥28 moderate to severe hot flushes/night sweats per week for 2 weeks before Visit 4 (week 0).
4. Subject is willing to maintain habitual diet (with the exception of restricted foods/beverages), physical activity patterns, and body weight during the study period.
5. Subject is willing to abstain from using products (other than study product) that contains estrogen, progestin, or progesterone within 30 d prior to Visit 1 (week -3) and throughout the study trial.
6. If a smoker, subject is willing to maintain current smoking habits.
7. Subject has no health conditions that would prevent her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results.
8. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Subject has abnormal laboratory test results of clinical importance at Visit 1 (week -3) at the discretion of the Investigator.
2. Subject has a history or presence of clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, endocrine, hematologic, immunologic (including chronic inflammatory conditions), neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary disorders, that, in the opinion of the Clinical Investigator, could interfere with the interpretation of the study results.
3. Subject has a history or presence of any gastrointestinal condition that could potentially interfere with absorption of the study product (e.g., inflammatory bowel syndrome, celiac disease, history of gastric bypass surgery).
4. Subject has a history of estrogen-dependent neoplasia, atypical ductual hyperplasia of the breast, or undiagnosed vaginal bleeding.
5. Subject has a history of endometrial hyperplasia, melanoma, or uterine/endometrial breast or ovarian cancer.
6. Subject has uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at Visit 1 (week -3). One re-test will be allowed on a separate day for subjects whose blood pressure exceeds either of these cut points at Visit 1, in the judgment of the Clinical Investigator.
7. Subject has a history of any major trauma or major surgical event within two months of Visit 1 (week -3).
8. Subject has a history or presence of cancer in the prior 2 years to Visit 1 (week -3), except for non-melanoma skin cancer.
9. Subject has a contraindication to estrogen and/or progestin therapy or allergy/sensitivity to the use of estradiol and/or progesterone, soy, or any components in the study product.
10. Subject has used estrogen alone or estrogen/progestin, selective estrogen receptor modulator, testosterone, or estrogen/testosterone within 30 d prior to Visit 1 (week -3).
11. Subject has used any prescription or over-the-counter products/supplements (e.g., soy products, herbal supplements) that have potential to alter progesterone or estrogen activity or is being used to treat VMS within 30 d prior to Visit 1 (week -3).
12. Subject has self-described extreme or irregular dietary habits, in the opinion of the Clinical Investigator or has been diagnosed with an eating disorder.
13. Subject has elective hospitalizations planned (e.g., elective cosmetic procedures) during the study period.
14. Subject has been exposed to any non-registered drug product or has participated in another intervention study within 30 d prior to Visit 1 (week -3).
15. Subject has a recent history of (within 12 months of screening; Visit 1; week -3) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
16. Individual has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Vasomotor symptoms | [Time Frame: Change from baseline to Week 12]
  Daily frequency of vasomotor symptoms, including hot flushes and night sweats

SECONDARY OUTCOMES:
Vasomotor symptom | [Time Frame: Change from baseline to Weeks 4 and 8]
  Daily frequency of vasomotor symptoms, including hot flushes and night sweats
Hot Flush | [Time Frame: Change from baseline to Weeks 4, 8, and 12]
  Daily frequency of hot flush
Night Sweat | [Time Frame: Change from baseline to Weeks 4, 8, and 12]
  Daily frequency of night sweat
Vasomotor symptom severity - number | [Time Frame: Change from baseline to Weeks 4, 8, and 12]
  Average number of moderate-to-severe VMS episode per day
Vasomotor symptom severity - total score | [Time Frame: Change from baseline to Weeks 4, 8, and 12]
  Average of VMS severity total score
Hot flush symptom severity - number | [Time Frame: Change from baseline to Weeks 4, 8, and 12]
  Average number of moderate-to-severe hot flush episode per day
Hot flush severity - total score | [Time Frame: Change from baseline to Weeks 4, 8, and 12]
  Average of hot flush severity total score
Night sweat severity - number | [Time Frame: Change from baseline to Weeks 4, 8, and 12]
  Average number of moderate-to-severe night sweat episode per day
Night sweat severity - total score | [Time Frame: Change from baseline to Weeks 4, 8, and 12]
  Average night sweat severity total score
Insomnia score | [Time Frame: Change from baseline to Weeks 4, 8, and 12]
  Average insomnia score per day obtained from Insomnia severity questionnaire (ISIQ)
Sleep duration | [Time Frame: Change from baseline to Week 12]
  Average sleep duration per day, obtained from sleep tracker
Actual sleep duration | [Time Frame: Change from baseline to Week 12]
  Average actual sleep duration per day obtained from sleep tracker
Sleep efficiency | [Time Frame: Change from baseline to Week 12]
  Average sleep efficiency per day obtained from sleep tracker
Sleep onset latency | [Time Frame: Change from baseline to Week 12]
  Average sleep onset latency per day obtained from sleep tracker
Latency to persistent sleep | [Time Frame: Change from baseline to Week 12]
  Average latency to persistent sleep per day obtained from sleep tracker
Wake after sleep onset | [Time Frame: Change from baseline to Week 12]
  Average wake after sleep onset per day obtained from sleep tracker
Fatigue | [Time Frame: Change from baseline to Week 12]
  Average fatigue score obtained from Chalder fatigue scale. Higher scores mean a worse outcome.
Sleep quality | [Time Frame: Change from baseline to Weeks 4, 8, and 12]
  Average sleep quality obtained from Pittsburgh sleep quality index
Vaginal bothersome score | [Time Frame: Change from baseline to Week 12]
  Average bothersome score obtained from Vaginal bothersome symptoms diary
Vaginal aging score | [Time Frame: Change from baseline to Week 12]
  Average vaginal aging score obtained from Day-to-day impact vaginal aging questionnaire
Menopause-specific quality of life | [Time Frame: Change from baseline to Weeks 4, 8, and 12]
  Average score obtained from Menopause-specific quality of life
General quality of life | [Time Frame: Change from baseline to Week 12]
  Average score obtained from RAND-36 questionnaire
Mood | [Time Frame: Change from baseline to Weeks 4, 8, and 12]
  Average score obtained from Profile of mood states (POMS)

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No